CLINICAL TRIAL: NCT04836832
Title: A Phase Ib/II Study of Duvelisib and Acalabrutinib in Relapsed/Refractory Indolent Non-Hodgkin Lymphoma (DUAL Trial)
Brief Title: Acalabrutinib and Duvelisib for the Treatment of Relapsed/Refractory Indolent Non-Hodgkin Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decision
Sponsor: Narendranath Epperla (Other)
Responsible Party: Sponsor-Investigator, Narendranath Epperla, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20179; NCI-2021-01355 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-03-09; First posted 2021-04-08 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Nodal Marginal Zone Lymphoma; Recurrent Splenic Marginal Zone Lymphoma; Refractory Follicular Lymphoma; Refractory Indolent Non-Hodgkin Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Nodal Marginal Zone Lymphoma; Refractory Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — acalabrutinib; duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib, duvelisib) (Experimental): Patients receive acalabrutinib PO BID, and duvelisib PO BID on days 1-28. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 19, patients receive acalabrutinib PO BID for up to 60 months in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Drug: Duvelisib

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Drug: Duvelisib — Given PO
  Other Names: 8-Chloro-2-phenyl-3-((1S)-1-(7H-purin-6-ylamino)ethyl)isoquinolin-1(2H)-one; Copiktra; INK-1197; IPI-145

SUMMARY:
This phase Ib/II trial studies the side effects of acalabrutinib and duvelisib and how well they work in treating patients with indolent non-Hodgkin lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Acalabrutinib inhibits a signaling molecule called Bruton tyrosine kinase and blocks cancer cell proliferation, growth, and survival. Duvelisib is designed to block a protein called PI3 kinase in order to stop cancer growth and cause changes in the immune system that may allow the immune system to better act against cancer cells. Giving acalabrutinib and duvelisib together may work better to block cancer growth than therapy of either drug alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of acalabrutinib and duvelisib in patients with relapsed or refractory indolent non-Hodgkin lymphoma (iNHL).

II. Determine maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). III. To estimate the overall response rate (ORR, Lugano 2014, computed tomography [CT] based) of acalabrutinib in combination with duvelisib at 6 months in follicular lymphoma (FL) and marginal zone lymphoma (MZL) cohorts.

SECONDARY OBJECTIVES:

I. To evaluate the activity of acalabrutinib and duvelisib as measured by ORR based on positron emission tomography (PET) scan at 6 months, duration of response (DOR) and 2-year progression-free survival (PFS).

II. To capture patient-reported outcomes (PROs).

EXPLORATORY OBJECTIVE:

I. To determine the correlation of the clinical activity of acalabrutinib in combination with duvelisib with established biomarkers and identify putative novel markers.

OUTLINE: This is a phase Ib, dose-escalation study of duvelisib, followed by a phase II study.

Patients receive acalabrutinib orally (PO) twice daily (BID), and duvelisib PO BID on days 1-28. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 19, patients receive acalabrutinib PO BID for up to 60 months in absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Histologically confirmed iNHL of any of the following subtypes recognized by the World Health Organization (WHO) classification: follicular lymphoma and marginal zone lymphoma (splenic, nodal and extranodal)
* Patients must meet clinical criteria for requiring treatment
* At least two prior systemic therapies for FL (phase 2 portion) and one prior systemic therapy for MZL. Prior autologous stem cell transplant is permitted. Prior CAR-T cell therapy is permitted. For the phase 1 portion, patients receiving one prior systemic therapy are allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Creatinine clearance >= 50 ml/min using a 24-hour creatinine clearance or estimated creatinine clearance using the Cockcroft-Gault equation
* Bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 1.5 x ULN
* Absolute neutrophil count (ANC) > 1000/mm^3 (without growth factor support)
* Platelet > 75,000/mm^3 (without transfusion support)

  * Unless related to bone marrow involvement with the disease, in which case platelets must be > 50,000/mm^3
* Hemoglobin >= 8 gm/dL
* Willing and able to participate in all required evaluations and procedures in this study protocol
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information
* Radiographically measurable disease by computed tomography (CT) scan, defined as at least one node > 1.5 cm in size or assessable disease
* Woman of childbearing potential (WOCBP) who are sexually active must agree to use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib, and 30 days after the last dose of duvelisib. WOCBP should have negative pregnancy test at screening and follow up throughout the study. Male subjects must agree to use highly effective methods of contraception during the study and up to 1 month after last dose of duvelisib. Male fertility may be impaired based on animal data (per duvelisib label)

Exclusion Criteria:

* Prior exposure to a BCR inhibitor (e.g., BTK inhibitors, phosphoinositide-3 kinase [PI3K], or Syk inhibitors) or BCL-2 inhibitor
* Patients with grade 3B FL or clinical evidence of transformation to aggressive lymphoma
* Central nervous system (CNS) involvement
* Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer which will not limit survival to < 1 year
* Clinically significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Note: Subjects with controlled, asymptomatic atrial fibrillation can enroll in study
* Active bleeding or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura)
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* Prothrombin time (PT)/international normalized ratio (INR) or activated partial thromboplastin time (aPTT) (in the absence of lupus anticoagulant) > 2 x ULN
* Requires treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Note: Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug
* Major surgical procedure within 28 days of the first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Pregnancy or lactation, or intending to become pregnant during the study
* Concurrent participation in another therapeutic clinical trial
* Known history of infection with human immunodeficiency virus (HIV)
* History of progressive multifocal leukoencephalopathy
* Grade >= 2 toxicity (other than alopecia) continuing from prior anticancer therapy
* Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function
* Prior history of drug-induced colitis or drug-induced pneumonitis
* History of chronic liver disease or veno-occlusive disease
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine) or systemic steroids > 20 mg of prednisone (or equivalent) once daily (QD)
* Uncontrolled viral, bacterial, fungal or parasitic infection that is untreated or unresponsive to antimicrobial therapy

  * NOTE: Subjects on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met
* Concurrent administration of medications or foods that are strong or moderate inhibitors or strong inducers of cytochrome P450 3A (CYP3A). No prior use within 2 weeks before the start of study intervention
* Patients with prior allogeneic transplantation
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV) at screening
* History of tuberculosis treatment within the 2 years prior to study entry
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy). Subjects with clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea, vomiting or any other condition that will interfere significantly with drug absorption
* Active cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection (i.e., subjects with detectable viral load)
* Administration of a live or live attenuated vaccine within 6 weeks of study entry
* Infection with hepatitis B, hepatitis C

  * Subjects with a positive hepatitis B surface antigen (HBsAg)
  * Subjects with a positive hepatitis B core antibody (HBcAb) must have negative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) to be eligible and must be periodically monitored for HBV reactivation by institutional guidelines
  * Subject who are hepatitis C antibody (HepcAb) positive will need to have a negative polymerase chain reaction (PCR) and must be willing to undergo DNA PCR testing during the study to be eligible
  * Investigators who strongly believe that a positive HBcAb is false (negative hepatitis C [hep C] PCR) due to passive immunization from previous immunoglobulin infusion therapy should consider the risk-benefit for the patient given the potential for reactivation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after completion of treatment
  Adverse events and toxicities of the combination regimen will be summarized using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria; toxicities will be tabulated overall and also by dose level.
Overall response rate (ORR) (assessed by computed tomography) | At 6 months
  Will be defined as the proportion of patients achieving a complete or partial response according to the Lugano Lymphoma Response Criteria by 6 months; any eligible patient who begins treatment with the combination regimen will be included in the denominator when calculating the ORR. ORR will be reported with a 95% binomial exact confidence interval.

SECONDARY OUTCOMES:
Complete response (CR) (assessed by positron emission tomography) | At 6 months
  Will be defined as the proportion of patients achieving a complete response according to the Lugano Lymphoma Response Criteria by 6 months; any eligible patient who begins treatment with the combination regimen will be included in the denominator when calculating the CR. CR will be reported with a 95% binomial exact confidence interval.
Duration of response (DOR) | Time from the first tumor assessment supports the response to the time of confirmed disease progression or death due to any cause, whichever occurs first, assessed up to 60 months
  Will be estimated using Kaplan-Meier method. Approximate 95% confidence intervals (CIs) for median DOR will be computed using the formula proposed by Brookmeyer and Crowley.
Progression-free survival | Time from first dose to documented disease progression, or death from any cause, whichever occurs first, assessed at 2 years
  PFS rates at 2-year and 95% CIs will be estimated using Kaplan-Meier methodology. Median PFS and its 95% CI will be calculated.
Patient reported outcomes (PROs) | Up to 12 months
  This will be a descriptive outcome that will be reported cumulatively rather than individual domains. Measures and assessment points are as follows: Sociodemographics (Screening only), PRO-CTCAE and Mood (POMS-s) C1 thru 12-months (10 data points), Stress (IES) and Quality of Life (SF-36), C1 thru 12-months (4 data points), and Life Events, Social Network Index (SNI), and Anxiety (GAD-7) and Depressive (PHQ-9) symptoms (Screening/C1 and 12 months).

OTHER OUTCOMES:
Biomarker analyses | Up to 60 months
  The effect of acalabrutinib and duvelisib will be analyzed on blood and tissue (lymph node or bone marrow, if involved) samples. Correlations between subject characteristics and outcome measures and correlations among outcomes measures will be explored using regression models or other appropriate techniques.
Pharmacokinetics analyses | Up to 60 months
  Blood samples will be collected at baseline, after the first dose, and at a steady state for all the patients at each dose level during the phase 1 portion of the study. This will enable us to understand the impact that each study drug may have on the other at these time points.

CONTACTS AND LOCATIONS:
Overall Officials: Narendranath Epperla, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu